CLINICAL TRIAL: NCT00879619
Title: A Pilot Phase I/II Study to Evaluate the Effects of Taxotere/Prednisone Plus Sunitinib in Chemotherapy-Naïve, Hormone Refractory Prostate Cancer Patients With Biochemical Relapse
Brief Title: Taxotere/Prednisone Plus Sunitinib in Chemotherapy-Naïve, Hormone Refractory Prostate Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow accrual.
Sponsor: John P. Fruehauf (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, John P. Fruehauf, Dr. John P. Fruehauf, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 07-64; 2008-6187 (Other: University of California, Irvine); NCI-2010-00216 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-04-08; First posted 2009-04-10 (Estimated); Results first posted 2013-06-06 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer; Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sunitinib; Docetaxel; Prednisone; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy and enzyme inhibitor (Experimental): Patients receive docetaxel IV over 60 minutes on day 1, prednisone PO BID on days 1-21, and sunitinib malate PO QD on days 2-15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive sunitinib malate PO QD on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate; Drug: docetaxel; Drug: prednisone

INTERVENTIONS:
Drug: sunitinib malate — Given PO
  Other Names: SU11248; sunitinib
Drug: docetaxel — Given IV
  Other Names: TXT
Drug: prednisone — Given PO
  Other Names: Delta(1)-Cortisone; deltacortisone; deltadehydrocortisone; metacortandracin; PRD; PRED

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving docetaxel and prednisone together with sunitinib malate may kill more tumor cells.

PURPOSE: This pilot phase I/II trial studies the side effects and best way to give docetaxel and prednisone together with sunitinib malate and to see how well it works in treating patients with prostate cancer that progressed after hormone therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the response by prostate specific antigen (PSA) of docetaxel/prednisone plus sunitinib (sunitinib malate) in chemotherapy-naive, hormone refractory prostate cancer subjects with biochemical relapse.

SECONDARY OBJECTIVES:

I. To determine the objective response rate (ORR) and duration of response (DR) in subjects with measurable disease.

II. To determine overall survival (OS) and time to progression (TTP). III. To evaluate the safety and tolerability of sunitinib in combination with docetaxel and prednisone.

OUTLINE:

Patients receive docetaxel intravenously (IV) over 60 minutes on day 1, prednisone orally (PO) twice daily (BID) on days 1-21, and sunitinib malate PO once daily (QD) on days 2-15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients then receive sunitinib malate PO QD on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria

* Subjects must have a histological diagnosis of adenocarcinoma of the prostate
* Age ≥ 18
* Subjects must have metastatic prostate cancer deemed to be unresponsive or refractory to hormone therapy by one or more of the following (despite androgen deprivation and anti-androgen withdrawal when applicable) check all that apply.
* Subjects may have received prior surgery. However, at least 21 days must have elapsed since completion of surgery and Subject must have recovered from all side effects.
* Subjects must have adequate hepatic function as defined by:
* a serum bilirubin ≤1.5 x the institutional upper limit of normal (IULN),
* Serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamic-pyruvic transaminase (SGPT) ≤2.5 x the institutional upper limit of normal obtained within 14 days prior to start of therapy
* Subjects must have 2 pre-study PSA > 2ng/ml at least 1 week apart within 28 days prior to start of therapy
* Subjects must have been surgically or medically castrated. If method of castration is luteinizing hormone-releasing hormone (LHRH) agonist (leuprolide or goserelin), then the Subject should be willing to continue the use of LHRH agonists. Castration using LHRH agonist should not be interrupted and subjects who have stopped treatment should be willing to restart.
* Subjects must not take vitamins, herbs, or micronutrient supplement within 28 days prior to start of therapy.
* Prior external beam radiation therapy (to less than 30% of the bone marrow only) is allowed. This includes prior use of samarium, but subjects can not have received prior strontium. At least 28 days must have elapsed since the completion of radiation therapy and the Subject must have recovered from side effects. Soft tissue disease which has been radiated in the prior 2 months is not assessable as measurable disease.
* Subjects with a history of myocardial infarction are not eligible. Subjects must have a baseline EKG to rule out underlying cardiac disease within 42 days prior to registration. Subjects with a history of cardiac disease, specifically congestive heart failure (CHF) are ineligible unless their disease is well-controlled. Subjects with history of cardiovascular accident (CVA) or atrial fibrillation are ineligible.
* Subjects with a history of brain metastases or who currently have treated or untreated brain metastases are not eligible. Subjects with clinical evidence of brain metastases must have a brain CT or MRI negative for metastatic disease within 56 days prior to registration.

  *Liver function tests should be evaluated prior to each treatment.
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Subjects must have an adequate renal function as defined by:
* a serum creatinine ≤1.5 x the institutional upper limit of normal obtained within 14 days prior to start of therapy and a urine protein: creatinine (UPC) ratio of ≤ 1.0.
* Subjects must have the following hematological criteria (minimal values):
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin of ≥ 8.0gm/dL,
* White blood cell count ≥ 2500,
* Platelets ≥ 75,000/mm³
* Subjects must be able to take oral medications

Exclusion Criteria

* Subjects must not have received chemotherapy, biologic therapy or any other investigational drug for any reason within 28 days prior to start of therapy and must have recovered from toxicities of prior therapy to grade 1 or less with the exception of alopecia.
* Subjects may not have ongoing problems with bowel obstruction or short bowel syndrome characterized by grade 2 or greater diarrhea or malabsorptive disorders.
* Men of child bearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.
* Subjects with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 will be excluded
* Subjects should not have psychological, familial, sociological, or geographical conditions that do not permit medical follow-up or compliance with the study protocol.
* Subjects should not have any medical life-threatening complications of their malignancies
* Subjects should not have a known severe and/or uncontrolled concurrent medical disease (e.g., uncontrolled diabetes, uncontrolled chronic renal or liver disease, active uncontrolled infection, or HIV).
* Subjects should not have current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
* Baseline blood pressure of < or equal to 150/100 mmHg. Subjects with a blood pressure reading above this level should be initiated on anti-hypertensive therapy and may be considered for protocol treatment when their blood pressure is adequately controlled.
* Subjects with New York Heart Association (NYHA) Grade II or greater congestive heart failure are not eligible. Subjects must have a baseline multiple gated acquisition scan (MUGA) or Echocardiogram with a calculated ejection fraction > or equal to 50%.
* Subjects with clinically significant peripheral vascular disease are not eligible.
* Subjects with evidence of bleeding diathesis or coagulopathy are not eligible.
* Subjects with central nervous system or brain metastases are not eligible.
* Subjects who had major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study are not eligible.
* Subjects with minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 0 are not eligible.
* Subjects with history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess are not eligible.
* Subjects with serious, non-healing wound, ulcer, or bone fracture are not eligible.
* Subjects who are diagnosed of any other malignancy except non-melanomatous skin cancer in the past 5 years are not eligible.
* Subjects receiving anticoagulation therapy (e.g. Coumadin) prior to registration are not eligible. Subjects are permitted to have prior Coumadin for prophylaxis against agents that might produce blood clots. Subjects with low dose Aspirin (86mg) are acceptable.
* Subjects with active thrombophlebitis or hypercoagulability are not eligible. Subjects with known history of pulmonary embolus are not eligible.
* All Subjects must be informed and must sign and give written informed consent in accordance with institutional and federal guidelines. Subjects who are unable to comply with study and/or follow-up procedures are not eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-07; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Fruehauf, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Comprehensive Cancer Center, Orange, California, United States

REFERENCES:
- See also: (UCi Clinical Trials webpage — http://www.ucihs.uci.edu/cancer/clinical_trialsl.shtml

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date: July 2009 Primary completion date: October 2011 Study completion date: November 2011
Groups:
- Chemotherapy and Enzyme Inhibitor: Patients receive docetaxel IV over 60 minutes on day 1, prednisone PO BID on days 1-21, and sunitinib malate PO once daily (QD) on days 2-15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive sunitinib malate PO QD on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  prednisone : Given PO
  docetaxel : Given IV
  sunitinib malate : Given PO
Period: Overall Study
Arm/Group | Chemotherapy and Enzyme Inhibitor
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Chemotherapy and Enzyme Inhibitor: Patients receive docetaxel IV over 60 minutes on day 1, prednisone PO BID on days 1-21, and sunitinib malate PO QD on days 2-15. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients then receive sunitinib malate PO QD on days 1-28. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
  prednisone : Given PO
  docetaxel : Given IV
  sunitinib malate : Given PO
Arm/Group | Chemotherapy and Enzyme Inhibitor
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Prostate Specific Antigen (PSA) Response Rate
Description: Defined by >= 30% decline in PSA from baseline for at least 3 months during study entry. Response rates will be expressed with two-sided exact binomial confidence intervals. Significance of changes between pre- and after-treatment PSA or testosterone will be determined by the Wilcoxon signed-rank test. Associations between PSA response and tumor response will also be examined by Fisher's exact test.
Time Frame: Baseline, every 3 weeks, at study termination, and then for 3 years
Arm/Group | Chemotherapy and Enzyme Inhibitor
Number analyzed (Participants) | 0

2. Secondary Outcome: Rates of Tumor Response (ORR)
Description: Response rates will be expressed with two-sided exact binomial confidence intervals. The difference of response rates between different pre-treatment pathological stages or Gleason scores will also be examined by Fisher's exact test. Associations between PSA response and tumor response will also be examined by Fisher's exact test.
Time Frame: Every 2 months
Arm/Group | Chemotherapy and Enzyme Inhibitor
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DR)
Description: Response rates will be expressed with two-sided exact binomial confidence intervals.
Time Frame: Up to 3 years
Arm/Group | Chemotherapy and Enzyme Inhibitor
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Progression (TTP) by PSA Response and Disease Response
Description: Defined as an absolute increase in PSA of at least 2 ng/ml. For subjects with measurable disease, Response Evaluation Criteria In Solid Tumors (RECIST) criteria will be used. Significance of changes between pre- and after-treatment PSA or testosterone will be determined by the Wilcoxon signed-rank test. Associations between PSA response and tumor response will also be examined by Fisher's exact test.
Time Frame: Baseline, every 3 weeks, at study termination, and then for 3 years
Arm/Group | Chemotherapy and Enzyme Inhibitor
Number analyzed (Participants) | 0

5. Secondary Outcome: Survival
Description: Quantitative Kaplan-Meyer estimates of progression-free survival and overall survival will be determined.
Time Frame: At 2 and 3 years
Arm/Group | Chemotherapy and Enzyme Inhibitor
Number analyzed (Participants) | 0

6. Secondary Outcome: Qualitative and Quantitative Toxicity
Description: Severity will be categorized by toxicity grade according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events v3.0 (CTCAE). Categorical analysis of toxicities will be performed.
Time Frame: Every 3 weeks and at study termination
Arm/Group | Chemotherapy and Enzyme Inhibitor
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At first study drug treatment during the initial treatment period until 28 days after the last administration of study drug.
Arm/Group | Chemotherapy and Enzyme Inhibitor
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy and Enzyme Inhibitor (N=4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Subject went to the emergency department & admitted to ICU due to dehydration. Had low blood pressure & hydrated but developed aspiration pneumonia & sepsis symptoms. Treated with broad spectrum antibiotics & had cerebrovascular accident & intubated.

LIMITATIONS AND CAVEATS:
The study was terminated due to slow accrual. Zero subjects were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes